CLINICAL TRIAL: NCT00185380
Title: Multi-center, Open, Randomized, Dose Finding Phase II Study to Investigate Ultra Low Dose Levonorgestrel Contraceptive Intrauterine Systems (LCS) Releasing Different Amounts of Levonorgestrel Compared to MIRENA in Nulliparous and Parous Women in Need of Contraception.
Brief Title: Dose-finding Study for the Ultralow-dose Levonorgestrel Intrauterine Contraceptive System (LCS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 91412; 2004-002291-42 (EudraCT Number); 308901 (Other: Company internal)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2010-03-10 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-05

CONDITIONS: Contraception
MeSH Terms: interventions — Levonorgestrel

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- LCS12 (Experimental): Levonorgestrel intrauterine contraceptive system (LCS) releasing 12 microg/24h in vitro
  Interventions: Drug: Levonorgestrel IUS (BAY86-5028, G04209B)
- LCS16 (Experimental): Levonorgestrel intrauterine contraceptive system (LCS) releasing 16 microg/24h in vitro
  Interventions: Drug: Levonorgestrel IUS (BAY86-5028, G04209C)
- IUS20 (Mirena) (Active Comparator): Levonorgestrel intrauterine system (IUS) releasing 20 microg/24h in vitro
  Interventions: Drug: Levonorgestrel IUS (Mirena, BAY86-5028)

INTERVENTIONS:
Drug: Levonorgestrel IUS (BAY86-5028, G04209B) — Levonorgestrel intrauterine contraception system (IUS) releasing 12 microg/24 h in vitro, to be used for three years
  Arms: LCS12
Drug: Levonorgestrel IUS (BAY86-5028, G04209C) — Levonorgestrel intrauterine contraception system (IUS) releasing 16 microg/24 h in vitro, to be used for three years
  Arms: LCS16
Drug: Levonorgestrel IUS (Mirena, BAY86-5028) — Levonorgestrel Intrauterine contraception system (IUS) releasing 20 microg/24 h to be used for three years
  Arms: IUS20 (Mirena)

SUMMARY:
The purpose of this study is to investigate if drug doses lower than the one released from Mirena® would be as effective for contraception as Mirena®. Subjects participating in the study will be randomly assigned to be inserted with any of the three different intrauterine systems (IUSs). The IUSs are nearly alike except that the amount of hormone released from them is different.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.

Bayer Schering Pharma AG, Germany is the sponsor of the trial.

Although the title of the study describes "open", it was in fact single-blinded.

Issues on side effects are addressed in the Adverse Event section.

ELIGIBILITY:
Inclusion Criteria:

* Women with or without children and good general health and in need of contraception.
* Regular menstrual cycle without hormonal contraceptives.

Exclusion Criteria:

* Pregnant or lactating.
* Last delivery or abortion less than 12 weeks ago.
* Previous pregnancies outside the womb.
* Previous pelvic infections.
* Abnormal bleeding.
* Abnormal uterine cavity.
* Climacteric signs.
* Genital cancer.
* Liver diseases.
* Alcoholism or drug abuse.

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 742 (Actual)
Dates: Start 2005-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (31):
- Finland (10):
  - Espoo
  - Helsinki
  - Joensuu
  - Jyväskylä
  - Kotka
  - Kuopio
  - Lahti
  - Oulu
  - Tampere
  - Turku
- Hungary (4):
  - Békéscsaba
  - Eger
  - Nyíregyháza
  - Szeged
- Norway (6):
  - Drammen
  - Elverum
  - Kolbotn
  - Larvik
  - Oslo
  - Trondheim
- Sweden (8):
  - Gothenburg
  - Huddinge
  - Kalmar
  - Luleå
  - Norrköping
  - Örebro
  - Stockholm
  - Umeå
- United Kingdom (3):
  - Chesterfield, Derbyshire
  - Sheffield, South Yorkshire
  - Chesterfield

REFERENCES:
- [Result] Gemzell-Danielsson K, Schellschmidt I, Apter D. A randomized, phase II study describing the efficacy, bleeding profile, and safety of two low-dose levonorgestrel-releasing intrauterine contraceptive systems and Mirena. Fertil Steril. 2012 Mar;97(3):616-22.e1-3. doi: 10.1016/j.fertnstert.2011.12.003. Epub 2012 Jan 4. PMID 22222193
- [Result] Apter D, Gemzell-Danielsson K, Hauck B, Rosen K, Zurth C. Pharmacokinetics of two low-dose levonorgestrel-releasing intrauterine systems and effects on ovulation rate and cervical function: pooled analyses of phase II and III studies. Fertil Steril. 2014 Jun;101(6):1656-62.e1-4. doi: 10.1016/j.fertnstert.2014.03.004. Epub 2014 Apr 14. PMID 24726226

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Parous or nulliparous women in good general health and in need of contraception were recruited from medical clinics between April and Nov 2005.
Pre-assignment Details: Most screening failures were in-/exclusion criteria not met and over-screening. Randomized: 742 women, Treated: 738 women. Full analysis set (FAS), safety analysis set (SAF) and per protocol analysis set (PPS) were identical (738 subjects).
Period: Overall Study
Arm/Group | LCS12 | LCS16 | IUS20 (Mirena)
Started | 240 | 246 | 256
Subjects Received Treatment | 239 | 245 | 254
Completed | 174 | 174 | 182
Not Completed | 66 | 72 | 74
Not completed — Adverse Event | 41 | 43 | 48
Not completed — Lost to Follow-up | 0 | 4 | 3
Not completed — Pregnancy | 1 | 4 | 0
Not completed — Protocol Violation | 2 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 0
Not completed — Failed insertion | 1 | 1 | 2
Not completed — Planned pregnancy | 9 | 12 | 12
Not completed — No need for contraception | 3 | 3 | 3
Not completed — Could not attend visits | 2 | 0 | 4
Not completed — personal reason | 6 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LCS12 | LCS16 | IUS20 (Mirena) | Total
Number analyzed (Participants) | 239 | 245 | 254 | 738
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (5.44) | 32.1 (5.31) | 32.0 (5.21) | 32.1 (5.31)
Sex: Female, Male [Count of Participants; unit: Participants] — Whilst 742 subjects were randomized, only 738 were treated.
  Participants
    Female | 239 | 245 | 254 | 738
    Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pearl Index
Description: The Pearl Index (PI) is defined as the number of pregnancies per 100 woman years. The 3-year PI was obtained by dividing the number of pregnancies that occurred during the first three years of treatment by the time (in 100 women years) that the women were under risk of getting pregnant.
Time Frame: Up to 3 years
Population: All randomized women with a successful insertion were analyzed according to the treatment actually received and were included in the FAS, which was the set used for all safety and efficacy analyses. The PPS was identical to the FAS.
Measure: Median (95% Confidence Interval); unit: Number per 100 women years
Arm/Group | LCS12 | LCS16 | IUS20 (Mirena)
Number analyzed (Participants) | 239 | 245 | 254
Number per 100 women years | 0.17 [0.00 to 0.93] | 0.82 [0.27 to 1.92] | 0.00 [0.00 to 0.59]

2. Secondary Outcome: Number of Subjects With Total or Partial Expulsions
Description: The numbers of subjects with partial or total IUS expulsions (device displaced from its correct position within the uterus) were to be given by treatment.
Time Frame: Up to 3 years
Population: The analysis was performed on the FAS (all subjects who had an IUS inserted).
Measure: Number; unit: participants
Arm/Group | LCS12 | LCS16 | IUS20 (Mirena)
Number analyzed (Participants) | 239 | 245 | 254
participants
  total expulsion | 0 | 3 | 0
  partial expulsion | 1 | 2 | 4

3. Secondary Outcome: Bleeding Pattern by 90-day Reference Periods - Reference Period 1
Description: Subjects kept a bleeding diary and recorded any bleeding every day by category: none, spotting, light, normal or heavy. Any missing data were obtained by direct questioning.
Time Frame: day 1 to day 90
Population: The analysis was performed on the FAS (all subjects with an insertion) and included subjects with bleeding or spotting or both.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | LCS12 | LCS16 | IUS20 (Mirena)
Number analyzed (Participants) | 228 | 241 | 244
days
  Number of bleeding days (light, normal or heavy) | 15.1 (10.1) | 15.4 (12.2) | 14.3 (12.9)
  Number of bleeding/spotting days | 39.9 (18.7) | 39.2 (19.7) | 36.6 (19.8)
  Number of spotting only days | 24.8 (14.1) | 23.8 (12.9) | 22.2 (13.5)

4. Secondary Outcome: Bleeding Pattern by 90-day Reference Periods - Reference Period 2
Description: as for outcome 3
Time Frame: day 91 to day 180
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | LCS12 | LCS16 | IUS20 (Mirena)
Number analyzed (Participants) | 225 | 230 | 239
days
  Number of bleeding days (light, normal or heavy) | 8.2 (8.0) | 7.7 (8.0) | 7.6 (9.1)
  Number of bleeding/spotting days | 22.6 (14.3) | 21.8 (14.3) | 21.8 (16.8)
  Number of spotting only days | 14.4 (10.3) | 14.1 (9.8) | 14.2 (11.5)

5. Secondary Outcome: Bleeding Pattern by 90-day Reference Periods - Reference Period 3
Description: as for outcome 3
Time Frame: day 181 to day 270
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | LCS12 | LCS16 | IUS20 (Mirena)
Number analyzed (Participants) | 220 | 224 | 230
days
  Number of bleeding days (light, normal or heavy) | 6.4 (7.3) | 5.4 (6.9) | 5.3 (7.3)
  Number of bleeding/spotting days | 18.3 (12.9) | 16.7 (12.6) | 16.8 (14.2)
  Number of spotting only days | 12.0 (9.3) | 11.3 (8.4) | 11.5 (9.5)

6. Secondary Outcome: Bleeding Pattern by 90-day Reference Periods - Reference Period 4
Description: as for outcome 3
Time Frame: day 271 to day 360
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | LCS12 | LCS16 | IUS20 (Mirena)
Number analyzed (Participants) | 217 | 218 | 225
days
  Number of bleeding days (light, normal or heavy) | 5.5 (6.7) | 4.7 (6.4) | 4.2 (6.3)
  Number of bleeding/spotting days | 16.7 (11.4) | 15.0 (11.6) | 15.2 (12.3)
  Number of spotting only days | 11.2 (8.5) | 10.2 (7.9) | 11.0 (9.2)

7. Secondary Outcome: Bleeding Pattern by 90-day Reference Periods - Reference Period 12
Description: as for outcome 3
Time Frame: day 991 to day 1080
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | LCS12 | LCS16 | IUS20 (Mirena)
Number analyzed (Participants) | 165 | 169 | 178
days
  Number of bleeding days (light, normal or heavy) | 3.6 (6.0) | 3.0 (4.5) | 1.9 (3.6)
  Number of bleeding/spotting days | 12.8 (10.7) | 10.6 (9.3) | 8.8 (8.6)
  Number of spotting only days | 9.2 (8.4) | 7.7 (6.9) | 6.9 (6.7)

ADVERSE EVENTS:
Description: An additional pregnancy was not recorded as an SAE.
Arm/Group | LCS12 | LCS16 | IUS20 (Mirena)
Serious Adverse Events (participants affected / at risk) | 12/239 | 12/245 | 16/254
Other Adverse Events (participants affected / at risk) | 187/239 | 198/245 | 218/254
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCS12 (N=239) | LCS16 (N=245) | IUS20 (Mirena) (N=254)
Goitre (Endocrine disorders) | 1 | 0 | 0
Blindness unilateral (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0
Hernia obstructive (General disorders) | 1 | 0 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 2
Cervicitis (Infections and infestations) | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0
Encephalitis herpes (Infections and infestations) | 0 | 0 | 1
Pelvic inflammatory disease (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Body temperature increased (Investigations) | 0 | 0 | 1
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Post-traumatic epilepsy (Nervous system disorders) | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 2 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 5
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Abdominal hernia repair (Surgical and medical procedures) | 1 | 0 | 0
Adhesiolysis (Surgical and medical procedures) | 1 | 0 | 0
Knee arthroplasty (Surgical and medical procedures) | 0 | 0 | 1
Mammoplasty (Surgical and medical procedures) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCS12 (N=239) | LCS16 (N=245) | IUS20 (Mirena) (N=254)
Abdominal distension (Gastrointestinal disorders) | 40 | 49 | 50
Abdominal pain (Gastrointestinal disorders) | 19 | 19 | 23
Nausea (Gastrointestinal disorders) | 18 | 20 | 22
Abdominal pain lower (Gastrointestinal disorders) | 16 | 19 | 21
Oedema (General disorders) | 15 | 21 | 19
Vulvovaginal candidiasis (Infections and infestations) | 23 | 30 | 21
Sinusitis (Infections and infestations) | 16 | 20 | 22
Influenza (Infections and infestations) | 14 | 22 | 20
Urinary tract infection (Infections and infestations) | 22 | 18 | 13
Vaginal infection (Infections and infestations) | 14 | 11 | 21
Nasopharyngitis (Infections and infestations) | 14 | 13 | 18
Bronchitis (Infections and infestations) | 8 | 7 | 16
Vaginitis bacterial (Infections and infestations) | 12 | 9 | 8
Procedural pain (Injury, poisoning and procedural complications) | 18 | 21 | 24
Weight increased (Investigations) | 38 | 39 | 31
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 14 | 23
Headache (Nervous system disorders) | 63 | 63 | 82
Mood altered (Psychiatric disorders) | 43 | 30 | 38
Depression (Psychiatric disorders) | 13 | 6 | 10
Breast discomfort (Reproductive system and breast disorders) | 52 | 51 | 62
Ovarian cyst (Reproductive system and breast disorders) | 21 | 24 | 60
Breast pain (Reproductive system and breast disorders) | 20 | 35 | 27
Dysmenorrhoea (Reproductive system and breast disorders) | 14 | 19 | 18
Acne (Skin and subcutaneous tissue disorders) | 64 | 61 | 73
Seborrhoea (Skin and subcutaneous tissue disorders) | 16 | 18 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor is interested in the publication of the results of every study. As some of the information concerning the study drug and the sponsor's development activities may be strictly confidential, any publication manuscript (including conference contributions, etc.) must first be reviewed by the sponsor before its submission or presentation.